CLINICAL TRIAL: NCT03925961
Title: Role of Pre-operative Counseling in the Surgical Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study expired in IRB.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00161974
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2020-09

CONDITIONS: Patient Education

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control arm (No Intervention): All subjects in the control arm will receive the current preoperative and post operative instructions.
- 'education booklet' arm (Experimental): All subjects in the 'education booklet' arm will receive the current standard Johns Hopkins Community Physicians Surgery packet and the Patient Information Booklet, specific to participants' surgery
  Interventions: Other: Preoperative education
- 'education booklet and preoperative' arm (Experimental): All subjects in the 'education booklet and preoperative' arm will receive the current standard Johns Hopkins Community Physicians Surgery packet and the Patient Information Booklet, specific to participants' surgery. Those subjects randomized to the 'education booklet and preoperative' arm will receive a pre-operative phone call by the research study's lead nurse, Catherine Davidson, approximately 1 week after participants enroll in the study. She will review pre-operative and post-operative guidelines pertinent to participants' operative as outlined in the patient information booklet. The amount of time (in minutes) that this phone call takes will be recorded in an excel file sheet.
  Interventions: Other: Preoperative education

INTERVENTIONS:
Other: Preoperative education — The intervention is focused around providing patients with educational information in the pre-operative setting and determine if this improves patients' surgical experience.
  Arms: 'education booklet and preoperative' arm; 'education booklet' arm

SUMMARY:
The study will seek to determine if surgical patients do better or the same if participants undergo pre-operative counseling for elective laparoscopic same day surgery. The study hypothesizes that patients who receive a pre-operative education booklet and a phone call from a surgical registered nurse, compared to the current standard of care, will have higher satisfaction with regard to participants' surgical experience, decrease in the number of post-operative phone calls, decrease in the number of opioid medications, and decrease in the number of emergency department visits. The importance of this study is to understand what surgical clinical practices can do in the pre-operative setting to enhance a surgical patient's recovery.

DETAILED DESCRIPTION:
In the last decade there has been an increasing focus on the patient's pre-operative, operative and post operative experience to help patient's in participants' recovery. For example, the surgical community has focused on pathways such as Enhanced Recovery After Surgery (ERAS), to improve patient's outcome and surgical experience. Despite this emphasis, little has been described in the literature as to how surgeons can improve a patient's experience by counseling participants on what participants can expect before, during, and after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* General surgical patients who will undergo same-day laparoscopic ventral hernia, inguinal hernia, and gallbladder surgery at Howard County General Hospital with the general surgery practice at Johns Hopkins Community Physicians.

Exclusion Criteria:

* Patients less than 18 years of age
* Adults who lack the capacity to consent
* Pregnant women
* Prisoners
* Non-English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Difference in patient satisfaction as assessed by a 10-point scale | 1 year
  The study will compare patient satisfaction scores between the three arms of the study groups to determine if there is a difference in patient satisfaction. It will be based on a scale of 1 to 10, 10 being the most satisfied and 1 being the least.

SECONDARY OUTCOMES:
Number of cases with post operative Wound Occurrence | 1 year
Number of post operative emergency department (ED) visits | 1 year
Number of cases with post operative respiratory occurrences | 1 year
Number of cases with post operative Urinary tract occurrences | 1 year
Number of cases with post operative central nervous system (CNS) occurrences | 1 year
Number of cases with post operative cardiac occurrences | 1 year
Number of cases with other unclassified post operative occurrences | 1 year
Number of cases with post operative Return to the OR within 30 days | 1 year
Number of cases with post operative Readmission | 1 year
Difference in time spent (in minutes) talking to patients on the phone | 1 year
  The study will assess if there is a difference in the amount of total time spent talking to patients over the phone.
Difference in post-operative number of opioid tablets used | 30 days
  The study will assess if there is a difference in the number of opioid tablets used at post operative day 30. For the purposes of this study, study patients will be discharged home with a prescription for oxycodone 5mg.

CONTACTS AND LOCATIONS:
Overall Officials: Hadley Wesson, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The Investigators will not make the individual participant data (IPD) available to other researchers.